CLINICAL TRIAL: NCT01958541
Title: A Brief Behavioral Sleep Intervention for Depression Among Military Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Ann Bernert, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22427; W81XWH-10-2-0178 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-04

CONDITIONS: Insomnia; Depression; Suicidal Ideation
Keywords: Sleep; Insomnia; Suicidal Symptoms; Suicidal Ideation; Military Veteran; Service Member; Depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Suicidal Ideation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Intervention I (Experimental): This non-medication group treatment (Sleep Intervention I) consists of four 90-minute sessions.
  Interventions: Behavioral: Sleep Intervention I
- Behavioral Intervention II (Active Comparator): This non-medication group treatment (Sleep Intervention II) consists of four 90-minute sessions.
  Interventions: Behavioral: Sleep Intervention II

INTERVENTIONS:
Behavioral: Sleep Intervention I — Insomnia-focused behavioral treatment (4 sessions).
  Arms: Behavioral Intervention I
Behavioral: Sleep Intervention II — Insomnia-focused behavioral treatment (4 sessions).
  Arms: Behavioral Intervention II

SUMMARY:
This study investigates the impact of brief behavioral insomnia treatment on depressive symptoms among military veterans.

ELIGIBILITY:
* Age 18 or older
* Veteran
* Insomnia Symptoms
* Depression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2013-03; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Suicidal Ideation | Change from Baseline in Suicidal Ideation at 7 weeks

SECONDARY OUTCOMES:
Insomnia Symptoms | Change from Baseline in Insomnia Symptoms at 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Bernert, Ph.D., Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Stanford University, Stanford, California